CLINICAL TRIAL: NCT01700075
Title: Comparative Physical and Chemical Study of the Mechanisms of Atherosclerosis With Development of Concept of Treatment and Prevention
Brief Title: Physical and Chemical Study of Atherosclerosis Mechanisms
Acronym: PCSAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nazarbayev University (Other)
Collaborators: Ministry of Health, Kazakhstan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0109RK000079
Record Dates: First submitted 2012-09-21; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Myocardial Infarction; Coronary Artery Diseases; Diabetes Mellitus, Type 2; Atherosclerosis of Femoral Artery
Keywords: atherosclerosis, development of concept, weight loss therapy
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment (Active Comparator): Lipidlowering: "Atorvastatin" (Liprimar) - 40mg per day. Antihypertensive: "Diroton" (Lisinopril, Gedeon Richter Ltd) - 10mg twice per day and "Ditiazem" (calcium bloker from the benthodiazepines, Lannacher, Austria) - 90mg per day.
  Antihyperglycemic drugs: biguanides "Metformin" - 0.5 g two or tree times per day, or "Exenatide" - 5-10 µg per day.
  Anti-inflammatory: "TromboACC" (acetylsalicylate acid) up to 2 g per day and/or "Clopidogrel" (thienopyridine class antiplatelet agent) - 75mg per day.
  Interventions: Drug: Conventional treatment
- Weight loss treatment (Experimental): Weight loss treatment by administering a healthy very low-calorie, low-fat vegetables and salt diet and includes an adjustment and modify eating behavior and increased physical activity.
  Interventions: Dietary Supplement: Weight loss treatment

INTERVENTIONS:
Drug: Conventional treatment — Lipidlowering: "Atorvastatin" (Liprimar) - 40mg per day. Antihypertensive: "Diroton" (Lisinopril, Gedeon Richter Ltd) - 10mg twice per day and "Ditiazem" (calcium bloker from the benthodiazepines, Lannacher, Austria) - 90mg per day.
  Antihyperglycemic drugs: biguanides "Metformin" - 0.5 g two or tree times per day, or "Exenatide" - 5-10 µg per day.
  Anti-inflammatory: "TromboACC" (acetylsalicylate acid) up to 2 g per day and/or "Clopidogrel" (thienopyridine class antiplatelet agent) - 75mg per day.
  Other Names: Pathogenetic and symptomatic treatment
  Arms: Conventional treatment
Dietary Supplement: Weight loss treatment — Weight loss treatment by administering a healthy very low-calorie, low-fat vegetables and salt diet and includes an adjustment and modify eating behavior and increased physical activity.
  Other Names: vegetable and salt diet
  Arms: Weight loss treatment

SUMMARY:
Study the mechanisms of atherosclerosis based on a comparative study of physical and chemical properties of lipid tissues at various localization with subsequent development of concept of treatment and prevention.

DETAILED DESCRIPTION:
The chemical and physical properties of different lipids of body. The clinical part of the work is a prospective randomized comparative controlled clinical trial of patients with atherosclerotic diseases.

Developed the concept of "limited biological resources" of the body based on the increase in the expenditure of energy reserves of the body, allowing a critical look at overweight.

The role of overweight in the development of atheromatous fat was revealed. The positive results from the weight loss in patients with atherosclerotic disease were drawn. Developed the metabolic concept of atherosclerosis associated with evolutionary aging and conversion of lipids in hard atherosclerotic fat.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent form
* dyslipidemia (HDL <1.0 mmol / l, triglycerides (TG) in plasma ≥ 1,7 mmol / l or cholesterol ≥ 5,6 mmol /l)
* waist circumference ≥ 94.0 cm in men or ≥ 80,0 cm in women,
* BP ≥140/95 mm Hg or a patient is taking antihypertensive medications,
* fasting glucose ≥ 6,1 mmol / l or the patient is taking hypoglycemic agents,
* the possibility of treatment for 6 months and follow-up for 1 year

Exclusion Criteria:

* Absence of consent form
* Non-compliance of patient to necessary recommendations.
* The presence of mental illness.
* Complete immobilization of a patient (paresis, and paralysis).

Ages: 26 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
full recovery from atherosclerotic diseases | for 12 months
  Regression of atherosclerosis plaque in vessel: imaging methods (GE Vivid 7 Ultrasound; GE Healthcare Worldwide USA, Michigan), and computed tomography scans (AG Siemens Somatom Emotion 6, Germany, Muenchen).
  Improvement of clinical condition: by measurement of clinical presence status.

SECONDARY OUTCOMES:
normalised laboratory and instrumental data | for 12 month
  Weight loss: Tanita-SC330S Body Composition Analyzer (Tanita Corp., Tokyo, Japan) including weight (kg), body mass index (BMI, kg/m2), body composition parameters, including as fat mass (in % of total body weight and total kg), visceral fat rating (units), fat free mass (kg), total body water (in % and kg), muscle mass (in % and kg), bone mass (in % and kg), metabolic age (years), basal metabolic rate (kcal per day), and bioimpedance (Ohms).
  Rate of blood circulation: Dopler Ultrasound (GE Healthcare Worldwide USA, Michigan).
  Bone density: bone densitometry (Lunar Achilles Express Ultrasound; GE Healthcare USA, Madison).
  Imaging of internal organs and blood vessel diameter: computed tomography scans (AG Siemens Somatom Emotion 6, Germany, Muenchen).
  General clinical study of blood and urine, liver and kidneys function tests, glucose and lipids levels.
  Clinical condition in dynamics: clinical presence status.

CONTACTS AND LOCATIONS:
Overall Officials: Kuat P Oshakbayev, MD, PhD, DsC, Principal Investigator — Scientisic research institute of cardiology and internal diseases
Locations (1):
- Scientific Research Institute of Cardiology and Internal Diseases, Almaty, Kazakhstan

REFERENCES:
- [Derived] Oshakbayev K, Dukenbayeva B, Otarbayev N, Togizbayeva G, Tabynbayev N, Gazaliyeva M, Idrisov A, Oshakbayev P. Weight loss therapy for clinical management of patients with some atherosclerotic diseases: a randomized clinical trial. Nutr J. 2015 Nov 25;14:120. doi: 10.1186/s12937-015-0108-y. PMID 26608649